CLINICAL TRIAL: NCT05635149
Title: Predictive Factors for Outcomes of Fruquintinib Plus Immunotherapy in Metastatic Colorectal Cancer：An Observational Cohort Study
Brief Title: Predictive Factors for Outcomes of Fruquintinib Plus Immunotherapy in Colorectal Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor
Other Study IDs: UNION00168
Record Dates: First submitted 2022-11-22; First posted 2022-12-02 (Actual); Last update posted 2022-12-02 (Actual); Status verified 2022-11

CONDITIONS: Colorectal Adenocarcinoma
MeSH Terms: interventions — Radiotherapy; Pharmaceutical Preparations; HMPL-013

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples Without DNA — Baseline feces of the enrolled patients was collected

GROUPS / COHORTS (2):
- Fruquintinib and anti-PD-1 plus radiotherapy: Fruquintinib is administrated as 4mg orally, once daily for 2 weeks on/1 week off.
  anti-PD-1 antibody is administrated as 200mg once every 3 weeks. Patients with isolated or localized metastasis will receive radiotherapy.
  Interventions: Radiation: radiotherapy
- Fruquintinib and anti-PD-1 alone: Fruquintinib is administrated as 4mg orally, once daily for 2 weeks on/1 week off.
  anti-PD-1 antibody is administrated as 200mg once every 3 weeks.

INTERVENTIONS:
Radiation: radiotherapy — In radiotherapy group, the modality of radiotherapy was conventional radiotherapy (CRT) or stereotactic body radiotherapy (SBRT) for cancer.
  Other Names: drug; Fruquintinib and anti-PD-1
  Groups: Fruquintinib and anti-PD-1 plus radiotherapy

SUMMARY:
This study was an observational cohort study to investigate the efficacy predictors of fuquinitinib combined with anti-PD-1 monoclonal antibody for third-line treatment and above in Chinese patients with advanced colorectal cancer.

DETAILED DESCRIPTION:
Patients with histologically confirmed metastatic or unresectable MSS/MSI-L/pMMR colorectal adenocarcinoma refractory to or intolerant of fluorouracil, oxaliplatin and irinotecan based systemic treatment, were enrolled in the study. All patients will receive a third line therapy with fruquintinib and anti-PD-1 antibody. Clinical and radiographic assessment will be performed regularly. Patients will be treated until disease progression, untolerable toxicity or withdrawal of consent.

ELIGIBILITY:
Inclusion Criteria:

* Signed the Informed Consent Form
* Ages: 18-75 Years (concluding 18 and 75 Years)
* Pathologically confirmed unresectable metastatic colorectal cancer
* Failure to 2st line therapy
* pMMR/MSS type
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Life expectancy greater than 3 months
* At least one measurable lesion (larger than 10 mm in diameter by spiral CT scan, larger than 20 mm in diameter by conventional CT scan) according to RECIST1.1
* Sufficient organ functions as follows (any blood transfusion or cell growth factor use within 14 days before enrollment is not allowed):

Absolute Neutrophil Count (ANC) ≥1.5×109/L Platelet Count of ≥175×109/L; Hemoglobin≥90g/L; Total Bilirubin (TBIL) ≤1.5 x ULN; ALT and /or AST<1.5 x ULN; If there is liver metastasis, then ALT and/or AST<3.0 x ULN; Serum Creatinine (SCr) ≤1.5×ULN; Endogenous creatinine clearance rate ≥50ml / min；

* Man and woman who childbearing potential agrees to use adequate contraception
* Willingness to provide enough tumor tissues for PD-L1 expression test

Exclusion Criteria:

* Patients could not obey the study protocol.
* Previous therapy with VEGFR Inhibitor or anti-PD-1 antibody.
* Other malignancy within 5 years prior to study enrolment, except for cervical carcinoma in situ, basal or squamous cell skin cancer.
* Known brain or CNS metastases.
* Patients with any active autoimmune disease or a documented history of autoimmune disease within 4 weeks prior to enrollment.
* Prior allogeneic bone marrow transplantation or prior solid organ transplantation.
* Uncontrolled malignant ascites.
* Clinically significant cardiovascular diseases, including but not limited to acute myocardial infarction, severe / unstable angina pectoris or coronary artery bypass grafting within 6 months before enrollment; Congestive heart failure, New York Heart Association (NYHA) grade > 2; ventricular arrhythmia requiring drug treatment; LVEF (left ventricular ejection fraction) < 50%.
* Known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients.
* Participation in another clinical trial with any experimental drug within 4 weeks prior to enrollment.
* Clinically significant electrolyte abnormalities judged by researchers.
* Systolic blood pressure > 140mmHg or diastolic blood pressure > 90mmHg regardless of any antihypertensive drugs.
* Poorly controlled diabetes before enrollment.
* Any factors that influence the usage of oral administration and patients cannot take fruquintinib orally.
* Active gastric and duodenal ulcer, ulcerative colitis or uncontrolled hemorrhage in GI, or other conditions that may cause GI bleeding and perforation as determined by the investigator.
* Patients with obvious evidence of bleeding tendency or medical history within 3 months before enrollment, hemoptysis or thromboembolism within 12 months.
* Active infection or serious infection that is uncontrolled by drug (NCI CTCAE v. 5.0 Grade ≥ 2).
* History of clinically significant hepatic disease, including hepatitis B virus (HBV) infection with HBV DNA positive (copies ≥1×104/ml or >2000IU/ml); known hepatitis C virus infection with HCV RNA positive (copies ≥1×103/ml).
* Persisting toxicity related to prior therapy (NCI CTCAE v. 5.0 Grade > 1).
* Pregnant or breastfeeding female patient.
* Receive blood transfusion, blood products and hematopoietic factors such as albumin and granulocyte colony stimulating factor (G-CSF) within 14 days prior to enrollment.
* Other severe acute or chronic medical conditions including metabolic disorder, physical examination or laboratory abnormalities that may increase the risk associated with study participation or study treatment administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study.
* Urinary protein ≥ ++, and the 24-hour urine protein quantification is greater than 1.0 g.
* Use of immunosuppressive medication, or systemic/local immunosuppressive corticosteroids for complication.
* Patients considered unsuitable for inclusion in this study by the investigator.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Chinese adults, both male and female, with histologically confirmed metastatic or unresectable MSS/MSI-L/pMMR colorectal adenocarcinoma refractory to or intolerant of fluorouracil, oxaliplatin and irinotecan based systemic treatment, were enrolled in the study. Demographic information (i.e., age and gender) was collected.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 1 year
  PFS is defined as the time from randomization to the first documented disease

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | from date of randomization until the date of progressive disease or EOT due to any cause, assessed up to 1 year
  ORR is defined as percentage of participants achieving assessed complete response (CR) and partial response (PR) by the investigator according to the RECIST 1.1.
Adverse Event (AEs) | from the date of first dose to the 30 days post the last dose
  Safety will be evaluated by incidence, severity and outcomes of adverse events (AEs) and categorized by severity in accordance with the NCI CTC AE Version 5.0.
Gut microbiome analysis | 16S ribosomal RNA (rRNA) sequencing for the baseline fecal samples of some patients
  To explore the association of gut microbiome and the efficacy of the treatment

OTHER OUTCOMES:
Exploratory endpoint | from date of randomization until the date of progressive disease or EOT due to any cause, assessed up to 1 year
  To identify the correlation between PD-L1 expression and inflammatory factor score with clinical outcomes

CONTACTS AND LOCATIONS:
Locations (1):
- Min Jin, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No
The datasets will be presented in online repositories: National Center for Biotechnology Information (NCBI), Sequence Read Archive (SRA).

REFERENCES:
- [Derived] Cheng M, Jin M, Yang S, Zhao L, Yu D, Lin Z, Li P, Huang C, Liu J, Wang J, Xue J, Ma H, Hu J, Yang K, Zhang T, Liu H. Effect of radiotherapy exposure on fruquintinib plus sintilimab treatment in refractory microsatellite stable metastatic colorectal cancer: a prospective observation study. J Immunother Cancer. 2025 Jan 4;13(1):e009415. doi: 10.1136/jitc-2024-009415. PMID 39755582